CLINICAL TRIAL: NCT03007888
Title: A Randomized, Multiple Dose Study to Assess the Pharmacokinetics and Pharmacodynamics of IPX203 in Subjects With Advanced Parkinson's Disease
Brief Title: A Study to Assess the PK and Pharmacodynamics of IPX203 in Subjects With Advanced Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Impax Laboratories, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IPX203-B16-01
Record Dates: First submitted 2016-12-06; First posted 2017-01-02 (Estimated); Results first posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-02

CONDITIONS: Advanced Parkinson's Disease
Keywords: IPX203 (carbidopa-levodopa) Extended-Release capsules
MeSH Terms: interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IPX203 then Sinemet (Experimental): Participants first received IPX203 ER CD-LD Capsules for 15 days After a Washout Period of 7 days; participants then received Sinemet (IR CD-LD) Tablet for 15 days Study drug doses were determined based on the subject's prestudy IR CD-LD regimen The typical IPX203 dosing regimen was 3 times a day, dosed approximately every 7 to 8 hours.
  Interventions: Drug: Sinemet; Drug: IPX203
- Sinemet then IPX203 (Experimental): Participants first received Sinemet Capsules for 15 days After a Washout Period of 7 days; participants then received IPX203 ER CD-LD Capsules for 15 days Study drug doses were determined based on the subject's prestudy IR CD-LD regimen The typical IPX203 dosing regimen was 3 times a day, dosed approximately every 7 to 8 hours.
  Interventions: Drug: Sinemet; Drug: IPX203

INTERVENTIONS:
Drug: Sinemet — Immediate Release Tablet containing carbidopa-levodopa flexible dosing
  Other Names: IR CD-LD Tablets
Drug: IPX203 — Extended Release capsules containing carbidopa-levodopa flexible dosing
  Other Names: IPX203 ER CD-LD Capsules

SUMMARY:
Primary Objective:

To compare the pharmacokinetics (PK) of single and multiple doses of IPX203 with Immediate release carbidopa-levodopa (IR CD-LD) in subjects with advanced Parkinson's disease (PD).

Secondary Objectives:

To compare the pharmacodynamics of single and multiple doses of IPX203 with IR CD-LD.

To compare the efficacy of IPX203 with IR CD-LD following multiple doses.

To evaluate the safety of IPX203.

DETAILED DESCRIPTION:
IPX203 is an investigational product containing CD-LD.

IPX203-B16-01 Study Design:

A randomized, open-label, rater-blinded, multicenter, 2-treatment, 2-period, multiple-dose crossover study.

Approximately 30 qualified IR CD-LD-experienced advanced PD subjects will be randomized.

The study duration will be approximately 8 weeks, including the screening period.

ELIGIBILITY:
Eligibility will be determined at screening and Visit 1 of the study.

Inclusion Criteria:

* Diagnosed with idiopathic PD at age ≥ 40 years who are being chronically treated with stable regimens of CD-LD but experiencing motor complications.
* Hoehn and Yahr Stages 2, 3, or 4
* Montreal Cognitive Assessment (MoCA) score ≥ 24 at Screening Visit in "on" state.
* For the 4 weeks prior to the Screening, the subject experiences daily "wearing-off" episodes with periods of bradykinesia and rigidity and experiences an "off" state upon awakening on most mornings by history.
* Responsive to CD-LD therapy and currently being treated on a stable regimen with CD-LD for at least 4 weeks prior to Visit 1
* Typically experiences an "on" response with the first dose of IR CD-LD of the day (by subject history).
* By history, efficacy of the first morning dose of IR CD-LD lasts less than 4 hours

Exclusion Criteria:

* History of medical conditions or of a prior surgical procedure that would interfere with LD absorption, such as gastrectomy or proximal small-bowel resection.
* Liver enzyme values ≥ 2.5 x the upper limit of normal; or history of severe hepatic impairment.
* History of drug or alcohol abuse within the 12 months prior to Screening.
* Received within 4 weeks of Visit 1 or planning to take during participation in the clinical study: any doses of a controlled-release (CR) LD apart from a single daily bedtime dose or any doses of Rytary, additional CD (eg, Lodosyn) or benserazide (eg, Serazide), or catechol-O-methyl transferase inhibitors (entacapone or tolcapone) or medications containing these inhibitors (Stalevo). Received within 4 weeks of Visit 1 or planning to take during participation in the clinical study: nonselective monoamine oxidase (MAO) inhibitors, apomorphine, or dopaminergic blocking agents including antiemetics.
* History of psychosis within the past 10 years.
* Treatment with any dopamine antagonist antipsychotics for the purposes of psychosis or bipolar disorder within the last 2 years.
* Based on clinical assessment, subject does not adequately comprehend the terminology needed to complete the PD Diary.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Impax Study Director, Study Director — Impax Laboratories, LLC
Locations (11):
- United States (11):
  - Investigator 110, Little Rock, Arkansas
  - Site 114, Little Rock, Arkansas
  - Investigator 106, Boca Raton, Florida
  - Investigator 112, Naples, Florida
  - Investigator 113, Port Charlotte, Florida
  - Site 108, Tampa, Florida
  - Investigator 101, Farmington Hills, Michigan
  - Site 103, Durham, North Carolina
  - Investigator 109, Cleveland, Ohio
  - Site 115, Kirkland, Washington
  - Investigator 104, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 39 subjects were screened at 10 study sites between November 8, 2016 and August 1, 2017
Pre-assignment Details: 28 of 39 subjects were enrolled and randomized
Groups:
- IPX203 First Then Sinemet: Participants first received IPX203 ER CD-LD Capsules for 15 days After a Washout Period of 7 days; participants then received Sinemet (IR CD-LD) Tablets for 15 days Study drug doses were determined based on the subject's prestudy IR CD-LD regimen The typical IPX203 dosing regimen was 3 times a day, dosed approximately every 7 to 8 hours.
- Sinemet First Then IPX203: Participants first received Sinemet for 15 days After a Washout Period of 7 days; participants then received IPX203 for 15 days Study drug doses were determined based on the subject's prestudy IR CD-LD regimen The typical IPX203 dosing regimen was 3 times a day, dosed approximately every 7 to 8 hours.
Period: First Intervention (14 Days)
Arm/Group | IPX203 First Then Sinemet | Sinemet First Then IPX203
Started | 15 | 13
Completed | 14 | 13
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Washout (7 Days)
Arm/Group | IPX203 First Then Sinemet | Sinemet First Then IPX203
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0
Period: Second Interventions (14 Days)
Arm/Group | IPX203 First Then Sinemet | Sinemet First Then IPX203
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects who were enrolled and randomized to 1 of 2 treatment sequences
Groups:
- All Study Participants: The recommended first morning dose of IPX203 on Day 1 was based on the subject's prestudy IR CD-LD morning dose
  The initial IR CD-LD dosing regimen was the same as the subject's stable prestudy regimen (unless s/he was taking a single daily bedtime dose of CR CD-LD, either alone or in combination with IR CD-LD, in which case, the CR CD-LD dose was discontinued and substituted with a 1:1 milligram-equivalent IR CD-LD dose).
Arm/Group | All Study Participants
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.43 (10.057)
Sex: Female, Male [Count of Participants; unit: Participants]
  Gender: Female | 12
  Gender: Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 26
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28
Age at Parkinson's disease onset [Mean (Standard Deviation); unit: years] | 58.9 (11.8)
Duration of Parkinson's disease [Mean (Standard Deviation); unit: years] | 7.5 (4.8)
Hoehn and Yahr Score [Count of Participants; unit: Participants] — 0:Asymptomatic
  1. Unilateral involvement only
  2. Bilateral involvement without impairment of balance
  3. Mild to moderate involvement; some postural instability but physically independent; needs assistance to recover from pull test
  4. Severe disability; still able to walk or stand unassisted
  5. Wheelchair bound or bedridden unless aided
  Participants
    I | 0
    II | 24
    III | 4
    IV | 0
Montreal Cognitive Assessment Score (On State) [Count of Participants; unit: Participants] — The Montreal Cognitive Assessment (MoCA) was designed as a rapid screening instrument for mild cognitive dysfunction. it assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. Time to administer the MoCA is approximately 10 minutes. The total possible score is 0 to 30 points; a score of 26 or above is considered normal.
  Montreal Cognitive Assessment (MoCA) score ≥ 24 is required at Screening Visit in "on" state.
  Participants
    MoCA score<24 | 0
    MoCA score 24 to <26 | 3
    MoCA score 26 to <28 | 13
    MoCA score 28 to <30 | 7
    30 | 5
Movement Disorder Society version of the Unified Parkinson's Disease Rating Scale Part III while On [Mean (Standard Deviation); unit: units on a scale] — MDS-UPDRS Part III was administered pre-dose (baseline). It comprises 18 items (speech,facial expression,rigidity,finger tapping,hand movements,pronation-supination hand movements,toe tapping,leg agility,arising from chair,gait,freezing of gait,postural stability,posture,global spontaneity movement, postural tremor of hands,kinetic tremor of hands,rest tremor amplitude,constancy of rest tremor scored on a 5-point normal-to-severe scale including dyskinesia impact questions ranging from 0 to 90 points. The higher the score the more abnormality.
  units on a scale | 19.1 (6.4)
Movement Disorder Society version of the Unified Parkinson's Disease Rating Scale Part III while Off [Mean (Standard Deviation); unit: units on a scale] — MDS-UPDRS Part III was administered pre-dose (baseline). It comprises 18 items (speech,facial expression,rigidity,finger tapping,hand movements,pronation-supination hand movements,toe tapping,leg agility,arising from chair,gait,freezing of gait,postural stability,posture,global spontaneity movement, postural tremor of hands,kinetic tremor of hands,rest tremor amplitude,constancy of rest tremor scored on a 5-point normal-to-severe scale including dyskinesia impact questions ranging from 0 to 90 points. The higher the score the more abnormality.
  units on a scale | 42.5 (10.6)
Total "off" time from subject diary [Mean (Standard Deviation); unit: hours] | 5.2 (1.8)
Total Good "on" time from subject diary [Mean (Standard Deviation); unit: hours] | 9.9 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Levodopa Cmax Following First Dose on Day 1
Description: Single Dose predose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 5.5, 6, 6.5, 7, 7.5, and 8 hours postdose
Time Frame: Day 1
Population: Randomized subjects who completed both periods
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- IPX203: Participants who received IPX203 ER Capsules on Day 1 of the study
- Sinemet: Participants who received Sinemet (IR CD-LD) Capsules on Day 1 of the study
Arm/Group | IPX203 | Sinemet
Number analyzed (Participants) | 27 | 27
ng/mL | 2857.56 (1204.506) | 2173.30 (1240.774)

2. Primary Outcome: Levodopa Tmax Following First Dose on Day 1
Description: Single Dose predose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 5.5, 6, 6.5, 7, 7.5, and 8 hours postdose
Time Frame: Day 1
Population: Randomized subjects who completed both periods
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | IPX203 | Sinemet
Number analyzed (Participants) | 27 | 27
hour | 2.07 (0.997) | 0.94 (0.560)

3. Primary Outcome: Levodopa t1/2 Following First Dose on Day 1
Description: Single Dose predose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 5.5, 6, 6.5, 7, 7.5, and 8 hours postdose
Time Frame: Day 1
Population: Randomized subjects who completed both periods
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | IPX203 | Sinemet
Number analyzed (Participants) | 27 | 27
hour | 1.658 (0.4838) | 1.420 (0.3194)

4. Primary Outcome: Levodopa AUCt Following First Dose on Day 1
Description: Single Dose predose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 5.5, 6, 6.5, 7, 7.5, and 8 hours postdose
Time Frame: Day 1
Population: Randomized subjects who completed both periods
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | IPX203 | Sinemet
Number analyzed (Participants) | 27 | 27
ng.h/mL | 12107.60 (5793.881) | 3747.61 (1819.141)

5. Primary Outcome: Levodopa AUCinf Following First Dose on Day 1
Description: Single Dose predose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 5.5, 6, 6.5, 7, 7.5, and 8 hours postdose
Time Frame: Day 1
Population: Randomized subjects who completed both periods
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | IPX203 | Sinemet
Number analyzed (Participants) | 27 | 27
ng.h/mL | 13968.57 (7606.901) | 4308.37 (2123.057)

6. Primary Outcome: Levodopa Bioavailability Relative to IR CD/LD Following First Dose on Day 1
Description: Single Dose predose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 5.5, 6, 6.5, 7, 7.5, and 8 hours postdose
Time Frame: Day 1
Population: Randomized subjects who completed both periods
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | IPX203 | Sinemet
Number analyzed (Participants) | 27 | 27
Percentage | 88.965 (21.7583) | 0 (0)

7. Primary Outcome: Carbidopa Cmax Following First Dose on Day 1
Description: Single Dose predose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 5.5, 6, 6.5, 7, 7.5, and 8 hours postdose
Time Frame: Day 1
Population: Randomized subjects who completed both periods
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | IPX203 | Sinemet
Number analyzed (Participants) | 27 | 27
ng/mL | 500.35 (316.299) | 151.50 (103.225)

8. Primary Outcome: Carbidopa Tmax Following First Dose on Day 1
Description: Single Dose predose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 5.5, 6, 6.5, 7, 7.5, and 8 hours postdose
Time Frame: Day 1
Population: Randomized subjects who completed both periods
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | IPX203 | Sinemet
Number analyzed (Participants) | 27 | 27
hour | 2.61 (0.655) | 2.07 (0.675)

9. Primary Outcome: Carbidopa t1/2 Following First Dose on Day 1
Description: Single Dose predose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 5.5, 6, 6.5, 7, 7.5, and 8 hours postdose
Time Frame: Day 1
Population: Randomized subjects who completed both periods
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | IPX203 | Sinemet
Number analyzed (Participants) | 27 | 27
hour | 2.015 (0.5159) | 1.969 (0.7187)

10. Primary Outcome: Carbidopa AUCt Following First Dose on Day 1
Description: Single Dose predose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 5.5, 6, 6.5, 7, 7.5, and 8 hours postdose
Time Frame: Day 1
Population: Randomized subjects who completed both periods
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | IPX203 | Sinemet
Number analyzed (Participants) | 27 | 27
ng.h/mL | 1940.51 (1095.449) | 436.63 (286.286)

11. Primary Outcome: Carbidopa AUCinf Following First Dose on Day 1
Description: Single Dose predose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 5.5, 6, 6.5, 7, 7.5, and 8 hours postdose
Time Frame: Day 1
Population: Randomized subjects who completed both periods
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | IPX203 | Sinemet
Number analyzed (Participants) | 27 | 27
ng.h/mL | 2239.61 (1232.234) | 610.44 (407.305)

12. Primary Outcome: Carbidopa Bioavailability Relative to IR CD/LD Following First Dose on Day 1
Description: Single Dose predose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 5.5, 6, 6.5, 7, 7.5, and 8 hours postdose
Time Frame: Day 1
Population: Randomized subjects who completed both periods
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | IPX203 | Sinemet
Number analyzed (Participants) | 27 | 27
Percentage | 117.442 (43.4176) | 0 (0)

13. Primary Outcome: Levodopa Cmax Following First Dose on Day 15
Description: Multiple Dose predose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, and 10 hours postdose.
Time Frame: Day 15
Population: Randomized subjects who completed both periods
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- IPX203: Participant who receive IPX203 ER CD-LD Capsules on Day 15 of the study
- Sinemet: Participants who received Sinemet (IR CD-LD) on Day 15 of the study
Arm/Group | IPX203 | Sinemet
Number analyzed (Participants) | 27 | 27
ng/mL | 2767.96 (1258.525) | 2356.85 (1178.628)

14. Primary Outcome: Levodopa Tmax Following First Dose on Day 15
Description: Multiple Dose predose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, and 10 hours postdose.
Time Frame: Day 15
Population: Randomized subjects who completed both periods
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | IPX203 | Sinemet
Number analyzed (Participants) | 27 | 27
hour | 1.91 (1.241) | 0.83 (0.439)

15. Primary Outcome: Levodopa AUCtau Following First Dose on Day 15
Description: Multiple Dose predose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, and 10 hours postdose.
Time Frame: Day 15
Population: Randomized subjects who completed both periods
Measure: Mean (Standard Deviation); unit: ng.h/ML
Arm/Group | IPX203 | Sinemet
Number analyzed (Participants) | 27 | 27
ng.h/ML | 11213.76 (4887.246) | 3879.39 (1744.328)

16. Primary Outcome: Carbidopa Cmax Following First Dose on Day 15
Description: Multiple Dose predose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, and 10 hours postdose.
Time Frame: Day 15
Population: Randomized subjects who completed both periods
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | IPX203 | Sinemet
Number analyzed (Participants) | 27 | 27
ng/mL | 478.66 (290.584) | 145.67 (82.541)

17. Primary Outcome: Carbidopa Tmax Following First Dose on Day 15
Description: Multiple Dose predose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, and 10 hours postdose.
Time Frame: Day 15
Population: Randomized subjects who completed both periods
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | IPX203 | Sinemet
Number analyzed (Participants) | 27 | 27
hour | 2.52 (0.74) | 2.20 (0.639)

18. Primary Outcome: Carbidopa AUCtau Following First Dose on Day 15
Description: Multiple Dose predose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, and 10 hours postdose.
Time Frame: Day 15
Population: Randomized subjects who completed both periods
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | IPX203 | Sinemet
Number analyzed (Participants) | 27 | 27
ng.h/mL | 1892.39 (1017.537) | 415.83 (279.487)

ADVERSE EVENTS:
Time Frame: 15 days for each intervention plus 1 week washout up to a total of 37 days
Description: All 28 subjects received at least one dose of IPX203 and 27 subjects received at least one dose of IR CD-LD
Groups:
- IPX203: Participants received IPX203 ER CD-LD Capsules
- Sinemet: Participant received Sinemet (IR CD-LD) Tablets
- Washout Period: Washout between Period 1 and Period 2
Arm/Group | IPX203 | Sinemet | Washout Period
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/27 | 0/28
Serious Adverse Events (participants affected / at risk) | 1/28 | 0/27 | 1/28
Other Adverse Events (participants affected / at risk) | 10/28 | 2/27 | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IPX203 (N=28) | Sinemet (N=27) | Washout Period (N=28)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhorea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IPX203 (N=28) | Sinemet (N=27) | Washout Period (N=28)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratiory track infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 5 (5) | 0 (0) | 0 (0)
Dystonia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Occipital Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional State (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-10-05): https://cdn.clinicaltrials.gov/large-docs/88/NCT03007888/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/88/NCT03007888/SAP_001.pdf